CLINICAL TRIAL: NCT02787902
Title: Improving Communication and Collaboration for Weight Management in Mother-daughter
Brief Title: Weight Management in Mothers and Adult Daughters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Becky Marquez, Assistant Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 151345
Record Dates: First submitted 2016-02-22; First posted 2016-06-01 (Estimated); Last update posted 2021-10-12 (Actual); Status verified 2021-10

CONDITIONS: Overweight or Obese
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Communication (Experimental): Behavioral weight loss program with communication skills training
  Interventions: Behavioral: Communication
- Standard (Active Comparator): Standard behavioral weight loss program
  Interventions: Behavioral: Standard

INTERVENTIONS:
Behavioral: Communication — Behavioral weight management program adapted for mother-daughter dyads with communication skills training
  Arms: Communication
Behavioral: Standard — Behavioral weight management program adapted for mother-daughter dyads without communication skills training
  Arms: Standard

SUMMARY:
The purpose of this study is to develop, implement, and evaluate a behavioral weight management intervention with a communication training component for Mexican-American women. The study has three specific aims.

Aim 1: Develop a behavioral weight loss intervention that modifies evidence-based behavioral weight loss treatment using results from formative data collected from Mexican-American mother-daughter dyads. The adapted intervention will focus on improving dyadic communication and collaboration for providing reciprocal support for healthy eating and physical activity behaviors.

Aim 2: Implement and evaluate a pilot weight management program adapted for mother-daughter dyads. Dyads will be randomly assigned to partner-based treatment with or without communication skills training.

Aim 3: Evaluate associations between changes in weight, weight-related behaviors, and psychosocial variables with changes in measures assessing interpersonal communication.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Body mass index of 25-50 kg/m2
* Mexican or Mexican-American

Exclusion Criteria:

* Pregnancy or plans to become pregnant in the next year
* 5% weight loss in the last 3 months
* History of bariatric surgery
* Serious medical condition or psychological disorder

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Weight change | 16 weeks
  Change in weight from baseline to post-intervention (16 weeks).

SECONDARY OUTCOMES:
Anthropometrics | baseline and post-intervention (16 weeks)
Blood pressure | baseline and post-intervention (16 weeks)
Communication | baseline and post-intervention (16 weeks)
Relationship factors (dyad, family, social networks) | baseline and post-intervention (16 weeks)
Psychosocial factors | baseline and post-intervention (16 weeks)
Eating behavior | baseline and post-intervention (16 weeks)
Physical activity | baseline and post-intervention (16 weeks)
Weight control behavior | baseline and post-intervention (16 weeks)
Treatment attendance and adherence | between baseline and post-intervention (16 weeks)

CONTACTS AND LOCATIONS:
Locations (1):
- University of California San Diego, La Jolla, California, United States